CLINICAL TRIAL: NCT00196118
Title: A Non-Randomized Prospective Study of IVC Filter Retrieval
Brief Title: Study of IVC Filter Retrieval With the Günther Tulip Vena Cava Filter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 04-507-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-12-11 (Estimated); Status verified 2007-12

CONDITIONS: Pulmonary Embolism; Venous Thromboembolism
Keywords: Pulmonary Embolism; Venous Thromboembolism; Inferior Vena Cava Filter; IVC; PE
MeSH Terms: conditions — Pulmonary Embolism; Venous Thromboembolism

INTERVENTIONS:
Device: Günther Tulip Vena Cava Filter

SUMMARY:
The purpose of this study is to test the hypothesis that the Günther Tulip Vena Cava Filter can be removed after a period of implantation, when implanted in patients for the prevention of pulmonary thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be considered at high risk for PE, but placement of a permanent IVC filter is not likely to be required.
* Patient must have a patent internal jugular vein.
* Patient has given informed consent.

Exclusion Criteria:

* Patient is less than 18 years.
* Patient has a pre-existing filter
* Patient had indications for a permanent filter at the time of the initial evaluation.
* Patient has uncontrollable coagulopathy.
* Patient has a short life expectancy < 6 months.
* Patient has metastatic malignancy.
* Patient has a vena cava diameter over 30 mm, measured by vena cava sizing catheters.
* Patient has a contrast allergy that cannot be adequately pre-medicated.
* Patient is at risk of septic embolism.
* Patient has sepsis.
* Patient has a hypersensitivity to any of the components of the GT filter, specifically cobalt, nickel, and chromium.
* Patient has impaired renal function (creatinine > 2.0).
* Patient is pregnant or planning to become pregnant within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2005-04; Study Completion 2007-07

PRIMARY OUTCOMES:
The rate of successful filter retrieval following implant.

SECONDARY OUTCOMES:
The rate of complications related to Inferior Vena Cava Filter use.

CONTACTS AND LOCATIONS:
Overall Officials: Bob Smouse, MD, Principal Investigator — Peoria Radiology Research & Education Foundation
Locations (17):
- United States (17):
  - Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Hospital of Miami, Inc.: Baptist Cardiac & Vascular Institute, Miami, Florida
  - Atlanta Medical Center, Atlanta, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spectrum Health Butterworth & Blodgett Campuses, Grand Rapids, Michigan
  - Oregon Health & Sciences University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Utah Valley Regional Medical Center Department of Radiology, Provo, Utah
  - LDS Hospital: Department of Radiology, Salt Lake City, Utah
  - INOVA Alexandria, Alexandria, Virginia